CLINICAL TRIAL: NCT04920851
Title: Comparison of Cytokine Hemadsorption as an Immunomodulator Therapy in Covid 19 Patients With and Without Bacterial Sepsis
Brief Title: Cytokine Hemadsorption in Covid 19 Patients With Bacterial Sepsis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Derince Training and Research Hospital (Other)
Responsible Party: Principal Investigator, İLKE KÜPELİ, ASSOC. PROF, Biruni University
Other Study IDs: BIRUNI 1
Record Dates: First submitted 2021-06-09; First posted 2021-06-10 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-06

CONDITIONS: INTERLEUKIN 6

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Covid with sepsis: Covid patient with sepsis
  Interventions: Device: cytokine hemadsorption
- covid without sepsis: Covid patient without sepsis
  Interventions: Device: cytokine hemadsorption

INTERVENTIONS:
Device: cytokine hemadsorption — to compare the laboratory and clinical results of cytokine hemadsorption as an immunomodulation therapy in COVID-19 ICU patients with or without sepsis.

SUMMARY:
In this retrospective study, we aimed to compare the laboratory and clinical results of cytokine hemadsorption as an immunomodulation therapy in COVID-19 ICU patients with or without sepsis.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 patients were the available data of laboratory diagnosis of COVID-19 (a positive throat swab nucleic acid test or positive serum COVID-19 specific antibody test),
* patients with COVID-19 induced sepsis was detection of bacterial agent in blood or tracheal culture

Exclusion Criteria:

* below 18 aged
* those who did not undergo hemoperfusion

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 23 COVID-19 patients were the available data of laboratory diagnosis of COVID-19 (a positive throat swab nucleic acid test or positive serum COVID-19 specific antibody test), and the criteria for patients with COVID-19 induced sepsis was detection of bacterial agent in blood or tracheal culture
Sampling Method: Non-Probability Sample
Enrollment: 23 (Estimated)
Dates: Start 2021-06-10 (Estimated); Primary Completion 2021-07-05 (Estimated); Study Completion 2021-07-20 (Estimated)

PRIMARY OUTCOMES:
interleukin 6 | 1 month
  level of interleukin 6

CONTACTS AND LOCATIONS:
Locations (1):
- Biruni University, Istanbul, Küçükçekmece, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Guan WJ, Ni ZY, Hu Y, Liang WH, Ou CQ, He JX, Liu L, Shan H, Lei CL, Hui DSC, Du B, Li LJ, Zeng G, Yuen KY, Chen RC, Tang CL, Wang T, Chen PY, Xiang J, Li SY, Wang JL, Liang ZJ, Peng YX, Wei L, Liu Y, Hu YH, Peng P, Wang JM, Liu JY, Chen Z, Li G, Zheng ZJ, Qiu SQ, Luo J, Ye CJ, Zhu SY, Zhong NS; China Medical Treatment Expert Group for Covid-19. Clinical Characteristics of Coronavirus Disease 2019 in China. N Engl J Med. 2020 Apr 30;382(18):1708-1720. doi: 10.1056/NEJMoa2002032. Epub 2020 Feb 28. PMID 32109013
- [Background] Yang X, Yu Y, Xu J, Shu H, Xia J, Liu H, Wu Y, Zhang L, Yu Z, Fang M, Yu T, Wang Y, Pan S, Zou X, Yuan S, Shang Y. Clinical course and outcomes of critically ill patients with SARS-CoV-2 pneumonia in Wuhan, China: a single-centered, retrospective, observational study. Lancet Respir Med. 2020 May;8(5):475-481. doi: 10.1016/S2213-2600(20)30079-5. Epub 2020 Feb 24. PMID 32105632
- [Result] Zhang W, Zhao Y, Zhang F, Wang Q, Li T, Liu Z, Wang J, Qin Y, Zhang X, Yan X, Zeng X, Zhang S. The use of anti-inflammatory drugs in the treatment of people with severe coronavirus disease 2019 (COVID-19): The Perspectives of clinical immunologists from China. Clin Immunol. 2020 May;214:108393. doi: 10.1016/j.clim.2020.108393. Epub 2020 Mar 25. PMID 32222466
- [Result] Esmaeili Vardanjani A, Ronco C, Rafiei H, Golitaleb M, Pishvaei MH, Mohammadi M. Early Hemoperfusion for Cytokine Removal May Contribute to Prevention of Intubation in Patients Infected with COVID-19. Blood Purif. 2021;50(2):257-260. doi: 10.1159/000509107. Epub 2020 Jun 26. PMID 32594085
- [Result] Houschyar KS, Pyles MN, Rein S, Nietzschmann I, Duscher D, Maan ZN, Weissenberg K, Philipps HM, Strauss C, Reichelt B, Siemers F. Continuous hemoadsorption with a cytokine adsorber during sepsis - a review of the literature. Int J Artif Organs. 2017 May 29;40(5):205-211. doi: 10.5301/ijao.5000591. Epub 2017 May 19. PMID 28525674